CLINICAL TRIAL: NCT02755090
Title: Nitrous Oxide Versus Intravenous Sedation for Anesthesia
Acronym: NOVIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Society of Family Planning (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Rameet Singh, Chief, Division of Family Planning, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: UNMHSC 16-101
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-07

CONDITIONS: Pregnancy Termination in Second Trimester
Keywords: nitrous; pain
MeSH Terms: conditions — Pain | interventions — Nitrous Oxide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrous oxide and IV saline (Experimental): Participants in the nitrous oxide group will receive a scented face mask through which nitrous oxide will be administered. The nitrous content of the gas will be titrated up by 20% every 5 breaths with a goal of 70% N2O/ 30% O2 as tolerated by the participant. This group will also receive saline through an IV. All participants will receive local anesthesia in the form of a paracervical block and ibuprofen pre-operatively.
  Interventions: Drug: Nitrous Oxide; Drug: IV Saline
- Standard Care (IV Sedation and Oxygen) (No Intervention): Within the IV sedation group, women will receive 100mcg fentanyl and 2mg midazolam at least two minutes prior to initiation of the procedure. This group will also receive 100% oxygen by a scented face mask. All participants will receive local anesthesia in the form of a paracervical block and ibuprofen pre-operatively.

INTERVENTIONS:
Drug: Nitrous Oxide — Participants in the nitrous oxide group will receive a scented face mask through which nitrous oxide will be administered. The nitrous content of the gas will be titrated up by 20% every 5 breaths with a goal of 70% N2O/ 30% O2 as tolerated by the participant. This group will also receive saline through an IV. All participants will receive local anesthesia in the form of a paracervical block and ibuprofen pre-operatively.
  Arms: Nitrous oxide and IV saline
Drug: IV Saline
  Arms: Nitrous oxide and IV saline

SUMMARY:
This study is a multi-site, double-blinded, randomized, non-inferiority clinical trial of inhaled nitrous oxide with oxygen (N2O/O2) versus intravenous (IV) sedation, with fentanyl and midazolam, for pain management in adult women having a pregnancy termination procedure between 12 and 16 weeks gestational age.

DETAILED DESCRIPTION:
This study will evaluate whether nitrous oxide is a feasible and acceptable alternative to IV sedation for pain management during early second trimester D&E. Primary endpoints will include maximum procedural pain using the visual analog scale (VAS) as well as satisfaction with anesthesia using the Iowa Satisfaction with Anesthesia Scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* pregnancy termination at gestational age of 12-16 weeks
* able to read and understand either English or Spanish
* able to obtain reliable post-procedure transportation

Exclusion Criteria:

* contraindications to outpatient pregnancy termination
* contraindications to nitrous oxide use (such as pernicious anemia, current treatment with bleomycin chemotherapy, active upper respiratory illness, or COPD)
* intrauterine fetal demise
* chronic narcotic use
* known adverse reaction to nitrous oxide, Fentanyl, or Versed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rameet Singh, MD, MPH, Principal Investigator — University of New Mexico Health Sciences Center
Locations (2):
- United States (2):
  - University of Colorado, Denver, Colorado
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico

REFERENCES:
- [Derived] Thaxton L, Pitotti J, Espey E, Teal S, Sheeder J, Singh RH. Nitrous Oxide Compared With Intravenous Sedation for Second-Trimester Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2018 Nov;132(5):1192-1197. doi: 10.1097/AOG.0000000000002915. PMID 30303904

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrous Oxide and IV Saline: Participants in the nitrous oxide group will receive a scented face mask through which nitrous oxide will be administered. The nitrous content of the gas will be titrated up by 20% every 5 breaths with a goal of 70% N2O/ 30% O2 as tolerated by the participant. This group will also receive saline through an IV. All participants will receive local anesthesia in the form of a paracervical block and ibuprofen pre-operatively.
  Nitrous Oxide: Participants in the nitrous oxide group will receive a scented face mask through which nitrous oxide will be administered. The nitrous content of the gas will be titrated up by 20% every 5 breaths with a goal of 70% N2O/ 30% O2 as tolerated by the participant. This group will also receive saline through an IV. All participants will receive local anesthesia in the form of a paracervical block and ibuprofen pre-operatively.
  IV Saline
- Standard Care Group (IV Sedation and Oxygen): Within the IV sedation group, women will receive 100mcg fentanyl and 2mg midazolam at least two minutes prior to initiation of the procedure. This group will also receive 100% oxygen by a scented face mask. All participants will receive local anesthesia in the form of a paracervical block and ibuprofen pre-operatively.
Period: Overall Study
Arm/Group | Nitrous Oxide and IV Saline | Standard Care Group (IV Sedation and Oxygen)
Started | 19 | 20
Completed | 18 | 20
Not Completed | 1 | 0
Not completed — equipment malfunction | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrous Oxide and IV Saline | Standard Care Group (IV Sedation and Oxygen) | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Full Range); unit: years] | 27.5 [19 to 40] | 26.8 [18 to 42] | 27.1 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 8 | 8 | 16
  Race: Black or African American | 4 | 0 | 4
  Race: American Indian/ Alaska Native | 1 | 3 | 4
  Race: Other: including bi and mutiracial | 6 | 9 | 15
Relationship Status [Count of Participants; unit: Participants]
  In a committed relationship | 13 | 13 | 26
  Not in a committed relationship | 6 | 7 | 13
Education [Count of Participants; unit: Participants]
  High school or equivalent | 8 | 8 | 16
  More than high school | 8 | 9 | 17
  Bachelor's or graduate degree | 3 | 3 | 6
Gestational Age [Count of Participants; unit: Participants]
  12 weeks | 8 | 8 | 16
  13 weeks | 3 | 4 | 7
  14 weeks | 5 | 5 | 10
  15 weeks | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Score for Maximum Procedural Pain
Description: To compare women's maximum procedural pain measured on a visual analog scale (VAS) during a surgical abortion between 12 weeks 0 days to 16 weeks 0 days gestational age between women randomized to nitrous oxide versus intravenous sedation. A score of 0 represents no pain and a score of 100 represents pain as bad as it could be.
Time Frame: Assessed immediately following completion of the procedure (as defined as removal of the speculum)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Nitrous Oxide and IV Saline | Standard Care Group (IV Sedation and Oxygen)
Number analyzed (Participants) | 18 | 20
units on a scale | 54.1 [40 to 68.1] | 34.0 [21.0 to 46.9]

2. Primary Outcome: Satisfaction With Anesthesia (Iowa Satisfaction With Anesthesia Scale [ISAS])
Description: The Iowa Satisfaction with Anesthesia Scale (ISAS) was given to women following a surgical abortion. The ISAS score is the mean of 11 responses to questions regarding satisfaction with anesthesia and has a score range of -3 (disagree strongly) to 3 (agree strongly).
Time Frame: Assessed 30 minutes after procedure completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide and IV Saline | Standard Care Group (IV Sedation and Oxygen)
Number analyzed (Participants) | 19 | 20
units on a scale | 0.7 (1.0) | 1.8 (1.0)

ADVERSE EVENTS:
Time Frame: Through the duration of the study, approximately one year.
Arm/Group | Nitrous Oxide and IV Saline | Standard Care Group (IV Sedation and Oxygen)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT02755090/Prot_SAP_000.pdf